CLINICAL TRIAL: NCT06469775
Title: Low Intensity Shock Wave Therapy for Men With Mild to Moderate Erectile Dysfunction
Brief Title: LiSWT for Men With Erectile Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institution unable to purchase machine to start study.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Danielle Velez Leitner, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2023002194
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LiSWT (Experimental): men receiving LiSWT
  Interventions: Device: Low intensity shock wave
- Control (Active Comparator): Standard of care: phosphodiesterase 5 inhibitor therapy, vacuum erectile device, constriction bands, intracorporal injections, penile implant.
  Interventions: Combination Product: Control

INTERVENTIONS:
Device: Low intensity shock wave — 6 sessions of low intensity shock wave therapy, applied in 15 minute appointments once weekly.
  Other Names: MoreNova
  Arms: LiSWT
Combination Product: Control — Standard of care treatment: phosphodiesterase 5 inhibitor therapy, vacuum erectile device, constriction bands, intracorporal injections, and penile implant.
  Arms: Control

SUMMARY:
The goal of this a clinical trial to investigate the effect of low-intensity shock wave therapy on patients with erectile function. The main questions it aims to answer are:

1. Can low-intensity shock wave therapy (LiSWT) to the penis improve male sexual health, particularly erectile function?
2. What is the optimal LiSWT protocol (number of shocks, energy delivered, timeline, etc) for initial and maintenance therapy?

Researchers will compare validated questionnaires on erectile function in men treated with LiSWT compared to men who receive standard of care to see if there is an improvement in erectile function with LiSWT.

Participants will be asked to complete questionnaires at each visit. Those who choose to undergo LiSWT will receive 6 sessions, once per week.

DETAILED DESCRIPTION:
Patients meeting inclusion criteria will be prospectively recruited from a single urological practice (Rutgers Urology, 125 Paterson St. Suite 4100, New Brunswick, NJ 08901) for this prospective study. They will be consented by a member of the research team within clinic. All consents and patient data will be stored in a HIPAA-compliant RedCap database. Patients who do not consent to LiSWT but want to participate in the study will be enrolled as a part of the Control group. These patients will also be recruited from a single urological practice as noted above, and consented by a member of the research team within clinic.

Patients who consent to the treatment arm will undergo LiSWT in clinic (typically up to 5,000 shocks per session, up to 6 weekly sessions), administered by study personnel with the MoreNova device (FDA-registered as a class 1 Therapeutic massager). Patients will be assessed for LiSWT complications and for erectile response with validated questionnaires at regular intervals: 1 month, 3 months, 6 months, and 1 year from LiSWT initiation. The patient's insurance will not be billed for the LiSWT sessions, but they will be billed for the follow-up visits. It is typical practice at Rutgers Urology to have any ED patients follow-up at these regular intervals when trialing alternative ED therapies, such as phosphodiesterase-5 inhibitors or intracavernosal injections. These will occur at regular clinic follow-up appointments, either via secure telehealth using the Epic electronic medical record platform or within the clinic. The Sexual Health Inventory for Men (SHIM) is a five-question, abbreviated, validated questionnaire derived from the International Index of Erectile Function questionnaire. It is widely used by urologists to evaluate efficacy of ED treatments. The Erection Hardness Score (EHS) is another tool often used to evaluate and monitor the severity of ED.

Study patients will be compared to control patients with ED who elect for standard therapies and/or lifestyle modifications instead of LiSWT for ED. These control patients will be matched in a 1:1 ratio to the study patients and matched to study patients by age, SHIM and EHS scores, and co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Male sex presenting with mild to severe erectile dysfunction for at least six months, as defined by SHIM score 1-21 and/or an EHS 0-3
* Age >18
* Ability to make independent decisions (sign own consent)

Exclusion Criteria:

* Men reliant on penile injections for erections
* Men with current penile implant
* Prisoners
* Current anticoagulant / anti-platelet therapy
* Adults who cannot make their own medical decisions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Health Inventory for Men (SHIM) | Performed at baseline, and then at each follow-up appointment (3, 6, 12, 24 months)
  The Sexual Health Inventory for Men (SHIM) is a five-question, abbreviated, validated questionnaire derived from the International Index of Erectile Function questionnaire. It is widely used by urologists to evaluate efficacy of ED treatments. It is graded on a scale of 1-25, with higher scores indicating no signs of erectile dysfunction.

SECONDARY OUTCOMES:
Erection Hardness Score | Performed at baseline, and then at each follow-up appointment (3, 6, 12, 24 months)
  The Erection Hardness Score (EHS) is another tool often used to evaluate and monitor the severity of ED. It is a four-point scale (1-4), with a score of 4 indicating a completely hard and fully rigid erection.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Velez Leitner, MD, Principal Investigator — Rutgers Health
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Zanaty F, Badawy A, Kotb H, Elsarfy F, Salman B. Efficacy and safety of low-intensity extracorporeal shock wave therapy versus on-demand tadalafil for erectile dysfunction. Arab J Urol. 2022 Jun 24;20(4):189-194. doi: 10.1080/2090598X.2022.2090134. eCollection 2022. PMID 36353469
- [Background] Yao H, Wang X, Liu H, Sun F, Tang G, Bao X, Wu J, Zhou Z, Ma J. Systematic Review and Meta-Analysis of 16 Randomized Controlled Trials of Clinical Outcomes of Low-Intensity Extracorporeal Shock Wave Therapy in Treating Erectile Dysfunction. Am J Mens Health. 2022 Mar-Apr;16(2):15579883221087532. doi: 10.1177/15579883221087532. PMID 35319291